CLINICAL TRIAL: NCT06427265
Title: Machine Learning-based Longitudinal Study of Post-ICU Syndrome Development Trajectory in Critically Ill Patients and Construction of Clinical Early Warning Models: a Research Protocol for Longitudinal Study
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital Of Guizhou Medical University (Other)
Collaborators: Chinese nursing association (Unknown)
Responsible Party: Sponsor
Other Study IDs: ZHKYQ202316; No. ZHKYQ202316 (Other Grant/Funding Number: Chinese Nursing Association); No. Gyfynsfc[2023]35 (Other Grant/Funding Number: The Affiliated Hospital of Guizhou Medical University)
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-06

CONDITIONS: Intensive Care Unit Syndrome; Prediction; Cognitive Impairment; Sleep Disorder; Memory Disorders
Keywords: Post-icu syndrome; Prediction model; Development Trajectory
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Wake Disorders; Memory Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project intends to track and evaluate whether post-ICU syndrome will occur 7 days, 1 month, 3 months and 6 months after ICU patients are transferred out of the ICU through a longitudinal study, apply the latent category growth model to identify different trajectory patterns of post-ICU syndrome in critically ill patients, and use modern machine learning models to build an early warning model of the trajectory patterns of post-ICU syndrome.

ELIGIBILITY:
Inclusion Criteria patients :

* Length of stay in ICU ≥24h;
* Age ≥18 years old;
* Conscious when leaving ICU, communicating with investigators without barriers;
* Informed consent. Family members：
* One family member ≥18 years of age was selected for each patient;
* Assume the main role of caring for patients and medical decision-making;
* No history of mental illness or other serious organic diseases;
* Informed consent and voluntary participation in this study.

Exclusion Criteria patients :

* Have been in ICU for more than 24h within 3 months before this admission;
* Transferred to another ICU;
* Cognitive impairment existed before ICU admission (BDRS > 4 points);
* Severe hearing impairment, dysarthria, etc., which cannot be followed up;
* Unable to complete the questionnaire survey due to serious illness.

Family members:

* Family members refuse to participate in the study due to their own reasons;
* Severe hearing and language impairment, unable to cooperate with researchers.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stage one involved studying patients discharged from the ICU and their families to investigate the occurrence and factors influencing post-intensive care syndrome (PICS), identifying various developmental patterns of PICS. A minimum sample size of 840 patients and 420 family members was established. Stage two focused on developing and evaluating a machine learning-based early warning model for PICS. The model construction utilized data from stage one, while the evaluation included 525 patients and 393 family members who met the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation scale score | 2024-2026
  Patient:
  1. Post-icu syndrome assessment of ICU survivors: Healthy Aging Brain Care monitoring(HABC Monitor) score;
  2. ICU related Memory: Intensive Care Unit Memory Tool (ICUMT);
  3. Sleep quality: Richards-Campbell Sleep Questionnaire (RCSQ);
  4. Perceived Social Support Scale (PSSS).
  Family members:
  1. Sleep quality of family members: Richards-Campbell Sleep Questionnaire (RCSQ);
  2. anxiety and Depression of family members: Hospital anxiety and Depression Scale score;
  3. Family fatigue: Scores of fatigue rating Scale;
  4. PTSD of family members: Event Impact Scale score;

CONTACTS AND LOCATIONS:
Overall Officials: Li Yao, Study Chair — Affiliated Hospital of Guizhou Medical University
Locations (1):
- Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No